CLINICAL TRIAL: NCT02917486
Title: EC-MOTION : ExtraCorporeal Membrane Oxygenation and Therapeutic Drug Monitoring of Drugs of infectION
Acronym: EC-MOTION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_8901
Record Dates: First submitted 2016-09-05; First posted 2016-09-28 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-08

CONDITIONS: Infection
Keywords: ExtraCorporeal Membrane Oxygenation; patient in intensive care; pharmacokinetic modeling
MeSH Terms: conditions — Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- ECMO piperacillin: patients in intensive care treated with ECMO with antiinfective therapy : piperacillin
  Interventions: Other: blood sample
- without ECMO piperacillin: patients in intensive care without ECMO with antiinfective therapy : piperacillin
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
The objective of the study is to investigate the exposure difference between antibiotic studied patients in intensive care with Extracorporeal Membrane Oxygenation and patients without Extracorporeal Membrane Oxygenation.

The exhibition is evaluated by population pharmacokinetic modeling.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Hospitalisation in intensive care
* Treatment with ECMO or without ECMO
* Introducing sepsis treated with an anti-infective molecule studied (piperacillin) for less than 48 hours
* With an arterial catheter
* Patient Information or their next of kin according to the patients status.

Exclusion Criteria:

* Pregnancy
* Major person under legal protection (backup justice, trusteeship, quardianship), person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in intensive care treated with ECMO or without ECMO
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Measure exposure to piperacillin | Day 1
  evaluated by population pharmacokinetic modeling and is defined by the time during which the antibiotic concentration is greater than 4 times the critical concentration of the germ to treat

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fillatre, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France